CLINICAL TRIAL: NCT04583254
Title: Hypofractionated External-beam RadiOtherapy for Intact Cervical Cancer (HEROICC-Trial): A Feasibility Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Principal Investigator, Lucas Mendez, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HEROICC; ReDA ID#10482 (Other: Lawson Health Research Institute)
Record Dates: First submitted 2020-10-02; First posted 2020-10-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cervical Cancer
Keywords: Hypofractionated External-beam Radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 EBRT+High-dose (HDR) Brachytherapy Experimental (Experimental)
  Interventions: Radiation: External beam radiotherapy (EBRT) + High-dose rate (HDR) Brachytherapy Experimental; Drug: Concurrent Chemotherapy
- Arm 2 EBRT+High-dose (HDR) Brachytherapy Standard of Care (Active Comparator)
  Interventions: Radiation: External beam radiotherapy (EBRT) + High-dose rate (HDR) Brachytherapy Standard of Care; Drug: Concurrent Chemotherapy

INTERVENTIONS:
Radiation: External beam radiotherapy (EBRT) + High-dose rate (HDR) Brachytherapy Experimental — 40 Gy / 15 Fractions EBRT + HDR-Brachytherapy
  Arms: Arm 1 EBRT+High-dose (HDR) Brachytherapy Experimental
Radiation: External beam radiotherapy (EBRT) + High-dose rate (HDR) Brachytherapy Standard of Care — 45 Gy / 25 Fractions EBRT + HDR-Brachytherapy
  Arms: Arm 2 EBRT+High-dose (HDR) Brachytherapy Standard of Care
Drug: Concurrent Chemotherapy — Weekly cisplatin 40 mg/m2 for a maximum of 5 cycles

SUMMARY:
External radiation given in 25 fractions or so together with weekly chemotherapy and followed by 3 or 4 fractions of brachytherapy is the standard of care for patients with locally advanced cervical cancer.

This study investigates the role of shortened external radiotherapy regimen (hypofractionated radiotherapy) by randomizing patients to this experimental regimen versus the standard of care.The purpose of this study is to access the feasibility of patient accrual to this trial in the Canadian setting and to provide an initial evaluation of cancer response and treatment tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* International Federation of Gynecology and Obstetrics (FIGO) IA or IB1 cervical cancers if not surgical candidates, but amenable to definitive chemoradiotherapy as proposed in this trial.
* FIGO Stage IB2, IB3, IIA or IIB cervical cancers
* FIGO stage IIIC1 cervical cancers are candidates but must meet all the following criteria:

  1. largest node is less than 3 cm
  2. less than 3 pathological nodes
  3. No nodes located in the common iliac chain.
  4. Cervical confined or with parametrial invasion
* Histologically-confirmed invasive uterine cervical carcinoma of subtypes squamous cell, adenocarcinoma or adenosquamous cell
* Candidate for definitive chemoradiotherapy to be delivered with weekly cisplatin
* Brachytherapy candidate

Exclusion Criteria:

* FIGO stage IIIA, IIIB, IIIC2, IVA or IVB
* FIGO stage IIIC1 with node greater than 3 cm, common iliac node or greater than 2 pathological nodes
* Previous pelvic or abdominal radiotherapy
* Patients requiring paraaortic nodal irradiation
* Inflammatory bowel disease
* Connective tissue disorder (eg. scleroderma, systemic lupus erythematous)
* Neuroendocrine, glassy cell, small cell, adenoid cystic carcinoma, adenoid basal carcinoma, clear cell, serous, endometrioid, verrucous carcinoma, melanoma, and sarcoma histologies
* Patient unable to undergo MR scan
* Eastern Cooperative Oncology Group (ECOG) performance status greater than 3
* Not a cisplatin candidate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-12-14 (Estimated); Study Completion 2028-12-14 (Estimated)

PRIMARY OUTCOMES:
Investigate the feasibility in the Canadian Health Care System | 3 years
  This trial aims to investigate its feasibility in the Canadian health care system. Feasibility will be defined as the ability to consent and randomize 48 patients over 3 years from date of site activation.

SECONDARY OUTCOMES:
Tumour response based on imaging | 3.5 years
  Tumour response rate on Magnetic resonance imaging (MRI) images will be graded as proposed in the EMBRACE 2 protocol

OTHER OUTCOMES:
Quality of Life (QoL) - Bowel and urinary quality of life as measured by the Expanded Prostate Cancer Index Composite (EPIC) questionnaire. | 8 years
  QoL will be measured by the Expanded Prostate Cancer Index Composite (EPIC) questionnaire. EPIC was initially created for assessment of QoL in patients with prostate cancers. This questionnaire was used in the NRG RTOG 1203 protocol (NCT01672892) and comprehensively assesses bowel function and bother (bowel summary domain) and urinary function, bother, incontinence and irritation/obstruction (urinary domain).
  The EPIC questionnaire contains 32 questions measuring patient function. Each question has a response option ranging from 0 or 1 (best) to 3, 4, or 5 (worst). The responses then correlate to a scoring scale of 0 to 100, where 0 is the best and 100 is the worst. The values vary from 0 to 100 for each question. The scores can then be added to come up with an overall quality of life score.
Quality of Life (QoL) is measured by European Organization for Research and Treatment of Cancer (EORTC) and Core 30 (QLQ-C30) QoL questionnaires | 8 years
  Two European Organization for Research and Treatment of Cancer (EORTC) QoL questionnaires (Core 30 (QLQ-C30). QLQ-C30 is used for all cancers and has several symptom scales, five functional scales (physical, emotional, social, role, cognitive) and a global health status scale.
  The QLQ-C30 responses are regarding function and symptoms are on a scale of 1 (not at all) to 4 (very much). Also included are questions about overall health and quality of life. Responses are on a scale of 1 (very poor) to 7 (excellent).
Quality of Life (QoL) - acute vaginal and sexual symptoms as measured by the cervical cancer module (QLQ-CX24) | 8 years
  QoL will be measured by the cervical cancer module (QLQ-CX24). QLQ-CX24 includes cancer - and treatment - related items and symptoms regarding sexuality. Acute and late vaginal and sexual QoL will be assessed using the QLQ-CX24 vaginal and sexual domains respectively.
  The QLQ-CX24 responses are regarding function and symptoms of sexual and vagina health. It is based on a scale of 1 (not at all) to 4 (very much).
Quality of Life (QoL) - late vaginal and sexual symptoms as measured by the cervical cancer module (QLQ-CX24) | 8 years
  QoL will be measured by the cervical cancer module (QLQ-CX24). QLQ-CX24 includes cancer - and treatment - related items and symptoms regarding sexuality. Acute and late vaginal and sexual QoL will be assessed using the QLQ-CX24 vaginal and sexual domains respectively.
  The QLQ-CX24 responses are regarding function and symptoms of sexual and vagina health. It is based on a scale of 1 (not at all) to 4 (very much).
Acute and late toxicity | 3 years and 3 months
  This outcome is assessed by physicians during each follow-up appointment, and scored according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (18). Clinically relevant toxicities of gastrointestinal, genitourinary, vaginal and non-specific general symptoms (i.e. fatigue, malaise and pain) will be collected. Hematological disorders will also be collected through weekly blood work checks. Acute toxicities will be collected at baseline, and then weekly during radiotherapy/chemoradiotherapy and at 3 months after completion of radiation. Late toxicities will be collected from 3 months after completion of radiation onwards until the end of follow-up.
Assessment of cancer down staging throughout EBRT. | 3 years
  To be assessed through volumetric comparison of gross tumor volume (GTV) and high risk clinical target volume (HR-CTV) contours in the pre-EBRT and brachytherapy MRI scans.
Progression-free survival | 8 years
  Defined as time from date of randomization to date of progression, date of death from any cause, or date of last follow-up, whichever occurs first. Cancer progression can be identified during physical exam, biopsy, or imaging of any kind.
Locoregional progression-free survival | 8 years
  Defined as time from date of randomization to date of locoregional progression, date of death from any cause, or date of last follow-up, whichever occurs first.
Metastasis-free survival | 8 years
  Defined as time from date of randomization to date of development of metastasis, date of death from any cause, or date of last follow-up, whichever occurs first.
Cervical cancer-specific survival | 8 years
  Defined as time from date of randomization to date of death attributed to cervical cancer, or date of last-follow-up, whichever occurs first.
Overall survival | 8 years
  Defined as time from date of randomization to date of death from any cause, or date of last follow-up, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas C Mendez, MD, Principal Investigator — London Health Sciences Centre, Lawson Health Research Institute
Locations (3):
- Canada (3):
  - BC Cancer - Kelowna, Kelowna, British Columbia
  - London Health Sciences Centre - London Regional Cancer Program, London, Ontario
  - Odette Cancer Centre - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No